CLINICAL TRIAL: NCT05667207
Title: Dipsticks and Point-of-care Microscopy to Reduce Antibiotic Use in Women With Uncomplicated Urinary Tract Infections: a Cluster-randomized Controlled Pilot Trial
Brief Title: Dipsticks and Microscopy to Reduce Antibiotic Use in Women's Urinary Tract Infections: a Pilot Trial (MicUTI)
Acronym: MicUTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital Erlangen (Other); LMU Klinikum (Other); University of Bristol (Other); University of Santiago de Compostela (Other); Università degli Studi di Trento (Other); University of Wuerzburg (Other); University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 109/22-sc
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2023-11

CONDITIONS: Cystitis Acute; Antibiotic Resistant Infection; Medication Adherence; Urinary Tract Infection Bacterial; Urinary Tract Infection Lower Acute
Keywords: General Practice; Primary care; randomized controlled trial; randomized clinical trial; cluster-randomized trial; pilot study; feasibility; microscopy; urinary dipsticks; clinical decision algorithm; point-of-care test
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Pilot study (feasibility)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care microscopy and dipstick guided management (Experimental): GPs whose practice is allocated to the intervention will have their management guided by POCTs, namely phase-contrast microscopy and urinary dipsticks for all patients consenting for participation.
  Interventions: Diagnostic Test: Point-of-care microscopy and dipstick guided management
- Usual care (No Intervention): Practices in the control arm will not have their management guided by POCTs. They will perform usual care. The treatment decision is usually based on symptoms and dip-stick test results (i.e., erythrocytes, leukocytes, nitrites).

INTERVENTIONS:
Diagnostic Test: Point-of-care microscopy and dipstick guided management — GPs will be encouraged to apply the following diagnosis and treatment algorithm (figure 1) to consenting women, taking their preferences into account:
  1. If POCTs are positive for bacteria by microscopy and/or for erythrocytes by dipsticks the GP issues, at his/her own clinical judgement, a delayed or immediate prescription for an antibiotic.10 In the MicUTI intervention, delayed prescription is defined as issuing an antibiotic prescription with the advice to take the medication only when symptoms do not improve or worsen in 48 hours.
  2. If POCTs are negative for bacteria and erythrocytes, the GP advises for self-help remedies according to guidelines and to do without antibiotics Study specific training in point-of-care microscopy will be provided to intervention practices.
  Arms: Point-of-care microscopy and dipstick guided management

SUMMARY:
With the aim to pilot a full-scaled trial to reduce unnecessary antibiotics in women with suspected uncomplicated urinary tract infections, twenty general practices in Bavaria, Germany, will be randomized to deliver patient management based on phase-contrast microscopy and urinary dipsticks or to usual care. Primary endpoints are recruitment and retention rates.

DETAILED DESCRIPTION:
Introduction: Uncomplicated urinary tract infections (UTIs) in women are among the most common infections encountered in primary care after those of the respiratory tract. They are often self-limiting, even though antibiotics are prescribed for almost all women presenting with suggestive clinical features. Efforts directed to tackle antimicrobial resistance led to primary care randomized controlled trials (RCTs) that investigated alternative treatment strategies in these patients. While reducing antibiotic use substantially, none of the experimental treatments showed non-inferiority to antibiotics with respect to clinical outcomes such as symptom duration, symptom burden, and pyelonephritis. Evidence suggests that rapid point-of-care (POC) tests to detect bacteria and erythrocytes in urine at presentation may help primary care clinicians to select women with uncomplicated UTIs (unUTIs) in whom antibiotics can be withheld without affecting clinical outcomes. The aim of this study is to pilot a full-scaled primary care RCT to evaluate the effects of a POC diagnosis and treatment algorithm based on a combination of phase-contrast microscopy and urinary dipsticks on antibiotic use in women with symptoms of an unUTI.

Methods and analysis: MicUTI (Microscopy in UTI) is a pragmatic open-label two -arm parallel pilot cluster-RCT. Twenty general practices affiliated to the Bavarian Practice Based Research Network (BayFoNet) in Germany will be randomly assigned to deliver patient management based on POC-tests (POCTs) or to the usual care arm. Urine samples will be obtained at presentation for POCTs and microbiological analysis. All patients will be followed-up using a self-directed patient diary completed until day 7 from inclusion or until symptom resolution (up to day 14), and through telephone-calls at day 28. An electronic medical record review is performed in case of missing follow-up information.

Primary endpoints are patient enrollment and retention rates. Exploratory endpoints include antibiotic use for UTI at day 28, time to symptom resolution, symptom burden, the number of recurrent and upper UTIs and re-consultations, and diagnostic accuracy (POCTs vs. urine culture as reference standard).

Ethics, data protection and trial registration: The trial will be conducted in accordance to the declaration of Helsinki and the relevant data protection regulations. Institutional review board approval: 109/22-sc (December 16, 2022)

ELIGIBILITY:
Inclusion Criteria:

* Women with at least two of dysuria, frequency, urgency, lower abdominal pain or hematuria.

Exclusion Criteria:

* Signs of a complicated UTI (anamnesis of fever, chills or flank pain)
* Clinically relevant immunosuppression (i.e., current use of any immunosup-pressive therapy, congenital or acquired disorders of immunity)
* Acute or chronic functional or anatomical variations in urinary tract except renal insufficiency grade II/IIIa
* Permanent bladder catheter or use of bladder catheter within the past two weeks
* UTI within the past two weeks
* Use of any antibiotic within the past two weeks
* Accommodation in a nursing home or hospital stay within the past two weeks
* Severe neurologic or psychiatric illness, severe dementia or severe substance use disorder
* Other severe diseases
* Being unable to understand the informed consent or to complete the patient diary
* Known pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment efficacy | 6 months (duration of the trial in each study site)
  Number of participants enrolled per site over 6 months of trial duration
Retention | 28 days (duration of the trial for each enrolled patient)
  Percentage of complete follow-ups over 28 days

SECONDARY OUTCOMES:
Total antibiotic use | 28 days
  Number of antibiotic prescriptions per patient with UTI within 28 days
Antibiotic doses | 28 days
  Defined daily doses of the prescribed antibiotics per patient with UTI within 28 days
Inappropriate antibiotic use | Day 0
  Percentage of patients with symptoms of UTI who were prescribed antibiotics among those with negative urine cultures
Immediate and delayed antibiotics | Day 0
  Number of immediate and delayed antibiotic prescriptions for uncomplicated UTI at initial consultation
Early relapses | Days 0-14
  Number of early relapses of UTI (days 0-14)
Recurrent urinary tract infections (UTIs) | Days 15-28
  Number of recurrent UTIs (day 15-28)
Upper UTIs | 28 days
  Number of upper UTIs within 28 days
Re-consultations | 28 days
  Number of consultations due to UTI (or symptoms of UTI) within 28 days
Symptom resolution | Days 0-7 (or max. 14 if symptoms last longer)
  Time to symptom resolution defined as a maximum of 1 point in each of the UTI-SIQ-8 items
Symptom Burden | Days 0-14
  Total symptom burden on days 0-7 (area under the curve of the UTI-SIQ-8 total symptom score)
Diagnostic accuracy | Day 0
  Diagnostic accuracy of microscopy +/- dipstick compared to the standard (urine culture)

CONTACTS AND LOCATIONS:
Overall Officials: Ildikó Gágyor, Professor, Principal Investigator — University Hospital Wuerzburg
Locations (2):
- Germany (2):
  - Stefanie Stark, Erlangen
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurotschka PK, Borgulya G, Bucher E, Endrich I, Figueiras A, Gensichen J, Hay AD, Hapfelmeier A, Kretzschmann C, Kurzai O, Lam TT, Massidda O, Sanftenberg L, Schmiemann G, Schneider A, Simmenroth A, Stark S, Warkentin L, Ebell MH, Gagyor I; Bavarian Practice-Based Research Network (BayFoNet). Dipsticks and point-of-care Microscopy to reduce antibiotic use in women with an uncomplicated Urinary Tract Infection (MicUTI): protocol of a randomised controlled pilot trial in primary care. BMJ Open. 2024 Mar 29;14(3):e079345. doi: 10.1136/bmjopen-2023-079345. PMID 38553055
- [Derived] Kurotschka PK, Koch MJ, Bucher E, Figueiras A, Gensichen J, Hapfelmeier A, Hay AD, Kretzschmann C, Kurzai O, Lam TT, Lasher K, Massidda O, Sanftenberg L, Schmiemann G, Schneider A, Simmenroth A, Stark S, Warkentin L, Ebell MH, Gagyor I; Bavarian Practice-Based Research Network (BayFoNet). Dipsticks and point-of-care Microscopy in Urinary Tract Infections in primary care: Results of the MicUTI pilot cluster randomised controlled trial. PLoS One. 2025 Oct 8;20(10):e0332390. doi: 10.1371/journal.pone.0332390. eCollection 2025. PMID 41060972
- [Derived] Sanftenberg L, Stofella J, Mayr K, Nassehi A, Hardtlein A, Stark S, Kuhlein T, Kurotschka PK, Gagyor I, Eck S, Schneider A, Bossenecker M, Roos M, Dreischulte T, Gensichen J; BayFoNet study group. Expectations of general practitioners on a practice based research network in Germany- a qualitative study within the Bavarian Research Practice Network (BayFoNet). BMC Prim Care. 2024 Jan 2;25(1):10. doi: 10.1186/s12875-023-02239-7. PMID 38166677
- [Derived] Sanftenberg L, Dreischulte T, Hardtlein A, Kosub H, Gagyor I, Kurotschka PK, Kuhlein T, Burggraf L, Eck S, Roos M, Gensichen J; BayFoNet-Research-Group. Process evaluation in practice based research networks: a study protocol for a mixed-methods implementation study. BMJ Open. 2023 Jul 12;13(7):e065947. doi: 10.1136/bmjopen-2022-065947. PMID 37438058
- See also: Study Protocol — https://bmjopen.bmj.com/content/14/3/e079345